CLINICAL TRIAL: NCT05697042
Title: A Mobile Intervention Merging Yoga and Self-Management Skills (MY-Skills Mobile) for Individuals Experiencing Symptoms of Long COVID-19
Brief Title: Merging Yoga and Self-Management Skills for Symptoms of Long COVID
Acronym: MYS LCOVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-2215
Record Dates: First submitted 2022-12-14; First posted 2023-01-25 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MY-Skills Mobile (Experimental): 8-week intervention merging yoga and self-management offered via secure remote tools including Zoom (video-conferencing software), Canvas (education software), and Qualtrics (survey software) that can be accessed via a computer or tablet. Each participant will have an initial yoga therapy individual session prior to start of group yoga. Group yoga is offered synchronously via Zoom two times per week for 60 minutes (120 minutes per week). The self-management content is delivered primarily through asynchronous tools that include educational videos, facilitated discussion boards, and interactive activities for goal setting, monitoring goals, and problem-solving practice. Self-management content is reiterated during the bi-weekly synchronous sessions, discussed as a group, and mantras are carried through both practices.
  Interventions: Behavioral: MY-Skills for Long COVID

INTERVENTIONS:
Behavioral: MY-Skills for Long COVID — 8 week online intervention with therapeutic yoga and self-management education

SUMMARY:
Long COVID patients experience high symptom burden for many months after initial infection of the COVID-19 virus. This study will investigate a mobile intervention Merging Yoga and Self-Management Skills (MY-Skills Mobile) as a complementary therapy for fatigue, pain, mood and quality of life in long COVID patients at the UCHealth Center for Integrative Medicine. The study aim is to assess the feasibility and acceptability of MY-Skills Mobile and research procedures including planned assessments.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the UC Health Integrated Medicine Clinic for long COVID
* community-dwelling
* speak English
* able to provide informed consent
* stand with or without an assistive device
* complete the Exercise Assessment and Screening for You (EASY) tool; potential participants will receive instructions about safe physical activity and/or to obtain physician approval prior to enrollment.

Participants will not be excluded due to limited technology access. We will loan tablets and hotspots to participants who do not have hardware or internet.

Exclusion Criteria:

* current yoga ≥120 minutes a week
* completed self-management education in the last year
* cognitive impairment limiting participation in decision making

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility- Recruitment | Week 1
  90% of screened patients will be eligible; 50% of eligible patients will consent
Feasibility- Use | Week 8
  >50% yoga session attendance and modules will be completed
Feasibility- Attrition | Week 8
  <20% attrition
Feasibility-Usability | Week 8
  User Mobile Application Rating Scale; <90% of participants to rate intervention between 3-5 (5-point scale)

SECONDARY OUTCOMES:
Symptom Burden Scale for Long COVID | Week 8
  Newly developed 14 scale for breathing, circulation, memory, thinking/communication, movement, sleep, ear/nose/throat, stomach, other symptoms and impact on daily life.
PROMIS Fatigue | Week 8
  13-item assessing fatigue experience and impact on function
Brief Pain Inventory | Week 8
  9-item for severity of pain and impact of pain on daily function
Short Form 36 | Week 8
  36-item function, pain, mental health, emotional well-being, fatigue, and general health perception

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Portz, PhD, MSW, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided